CLINICAL TRIAL: NCT05031286
Title: Differences in Sensitization Between Men and Women After Cutaneous Thermal Stimuli
Brief Title: Differences in Pain Processing Between Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Schweinhardt Petra, Head of Research at the Department of Chiropractic Medicine, Balgrist University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NWR
Record Dates: First submitted 2021-08-11; First posted 2021-09-01 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Central Sensitisation
Keywords: central sensitisation; central sensitization; nociception; withdrawal reflex; heat pain; secondary hyperalgesia
MeSH Terms: conditions — Hyperalgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Other: Cutaneous thermal stimuli

INTERVENTIONS:
Other: Cutaneous thermal stimuli — Application of thermal stimuli of different intensities to the skin

SUMMARY:
Many chronic pain conditions show clear differences between between men and women, such as reported pain intensities or treatment effects, with chronic pain conditions being generally more frequent in women. Yet, the underlying mechanisms causing these differences are poorly understood. Central sensitization (CS) is considered one important mechanism in pain patients which differs between female and male patients. The central hypothesis is that already in the healthy population CS processes are more pronounced in women than in men.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* able to give informed consent

Exclusion Criteria:

* pain complaints for more than two consecutive days over the past three months
* any major medical or psychiatric condition (e.g. heart disease, major depressive disorder)
* any chronic pain condition
* inability to follow study instructions
* consumption of stimulants, drugs, or analgesics within the past 24 hours
* scar tissue or generally reduced sensitivity in the designated testing site areas

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in spatial extent of mechanical hypersensitivity after intervention w.r.t. baseline | 10-20 minutes before intervention (baseline) and 20-30 minutes after intervention
  Mapping of hypersensitivity in cm2 of sensitized skin area using two quantitative sensory testing tools (256mN von Frey filament and 200-400mN brush) before and after intervention
Changes to the nociceptive withdrawal reflex (NWR) after intervention w.r.t. baseline | 5-10 minutes before intervention (baseline) and 30-35 minutes after intervention
  Repetitive suprathreshold elicitation of the NWR to monitor its characteristics (such as magnitude and number of responses) before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Petra Schweinhardt, MD, PhD, Principal Investigator — Department of Chiropractic Medicine, Balgrist University Hospital, University of Zurich
Locations (1):
- Balgrist Campus, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guekos A, Saxer J, Salinas Gallegos D, Schweinhardt P. Healthy women show more experimentally induced central sensitization compared with men. Pain. 2024 Jun 1;165(6):1413-1424. doi: 10.1097/j.pain.0000000000003144. Epub 2024 Jan 11. PMID 38231588